CLINICAL TRIAL: NCT03968562
Title: Assessment of Suppression of Cutaneous Allergic Responses and Pruritus by Topical Doxycycline
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: State University of New York - Downstate Medical Center (Other)
Responsible Party: Principal Investigator, Rauno Joks, MD, Chief Division of Allergy Immunology, State University of New York - Downstate Medical Center
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1349966
Record Dates: First submitted 2019-05-22; First posted 2019-05-30 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Hives
MeSH Terms: conditions — Urticaria

STUDY DESIGN:
Intervention Model Description: This cross-sectional survey involves a single consecutive two day study visit.To assess the effect of topical doxycycline 2% emollient cream or control emollient on immediate hypersensitivity allergy skin tests responses, pruritus, and associated late phase skin swelling. We will use generic Aquaphor, a skin protectant, as the control emollient. The active ingredient in this cream is Petrolatum 42%. Inactive ingredients include ceresin, lanolin alcohol, microcrystalline wax, mineral oil, phenoxyethanol. Adults (18-75 yrs) with known respiratory (allergic rhinoconjunctivitis and/or asthma), and are allergen skin prick test (SPT) positive to common aeroallergens will, after 5 days of non-use of oral antihistamine therapy, undergo limited repeat SPT with the same allergens (up to 5 allergens per subject) with measurement of swelling, flare, and itch at 20 min, then after application of doxycycline cream or control emollient, at 30 min, 60 min, and 24 hrs post initial cream removal.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 2% Doxycycline Cream in Generic Aquaphor (Active Comparator): 2% Doxycycline Cream in Generic Aquaphor will be applied topically twice during the study visit: first for 30 minutes, then for 6 hours duration. Will perform concurrent to Placebo Comparator
  Interventions: Drug: 2% Doxycycline Cream in Generic Aquaphor or Generic Aquaphor
- Generic Aquaphor (Placebo Comparator): Generic Aquaphor will be applied topically twice during the study visit: first for 30 minutes, then for 6 hours duration. Will perform concurrent to Active Comparator.
  Interventions: Drug: 2% Doxycycline Cream in Generic Aquaphor or Generic Aquaphor

INTERVENTIONS:
Drug: 2% Doxycycline Cream in Generic Aquaphor or Generic Aquaphor — 2% Doxycline Cream in Generic Aquaphor or Generic Aquaphor will be applied topically twice during the study visit: first for 30 minutes, then for 6 hours duration.

SUMMARY:
Investigators will study the effects of topical doxycycline on cutaneous allergic early and late phase responses by determining allergen skin responses in each subject after a single application to allergen induced allergic swelling of 2% doxycycline in emollient.

DETAILED DESCRIPTION:
This study is a cross-sectional survey to be completed in a single consecutive two day study visit.

To assess the effect of topical doxycycline 2% emollient cream or control emollient on immediate hypersensitivity allergy skin tests responses, pruritus, and associated late phase skin swelling.

Investigators will use generic Aquaphor, a skin protectant, as the control emollient. The active ingredient in this cream is Petrolatum 42%. Inactive ingredients include ceresin, lanolin alcohol, microcrystalline wax, mineral oil, phenoxyethanol.

Adults (ages 18-75 yrs) treated at the SUNY Downstate/UHB Allergy Faculty Practice with known respiratory (allergic rhinoconjunctivitis and/or asthma), and who have previously been evaluated and are allergen skin prick test (SPT) positive to common aeroallergens will, after five days of non-use of oral antihistamine therapy, undergo limited repeat SPT with the same documented positive allergens (up to 5 allergens per subject).

1. Allergen skin prick testing (Dermapik method) will be done on the volar surface of each forearm, with identical SPT allergens. The profile to be tested will be individualized, from 1-5- allergens, to be determined by previous skin test positive results. Volunteers for the study who have not been previously tested will also be eligible, provided they have a history of symptoms consistent with allergic rhinoconjunctivitis and/or asthma. These subjects will receive testing with a select panel of 5 mixed allergens - to include both perennial (cat, dust mite) and seasonal (tree, grass, ragweed).

   Each subject will also be tested with standardized negative and positive controls of saline and histamine. Two control sites, left and right mid upper back, will both be pricked with histamine and saline.
2. After 20 minutes, the initial baseline determination of mean diameter (average of widest and its orthogonal measurement) will be taken of both wheal and flare, as will itch scores for each arm and each back control site (VAS (0 to 100 mm line) and verbal rating scale ( 0 - none, 1 - mild, 2 - moderate, 4 - severe)).
3. The location (right versus left) of placement of medication (active) versus control will be determined by a random numbers list for both forearm and back evaluation test sites. The subject will be blinded as to identity of the cream applied at each site.

   Using a single blind approach, a thin film of either doxycycline 2% cream or control emollient will be placed on entire test surface of either arm for an additional 30 min then removed. Repeat skin and itch measurements will immediately be done.
4. After an additional 30 minutes after wiping off the cream repeat skin and itch measurements will be done.
5. Reapplication - Investigators will then apply repeat film of cream to allergen test surface sites only then send the subject home with instructions to not wash the sites off for 6 hrs.
6. Repeat measurements at 24 hours post initial removal of cream.

ELIGIBILITY:
Inclusion Criteria:

* Adult (ages 18-75) outpatients with diagnosis of allergic rhino-conjunctivitis and/or asthma who have previously undergone epicutaneous skin prick testing with detection of at least one allergen positive, and who may or may not have had a serum IgE level done as part of their routine evaluation.

Exclusion Criteria:

* Subjects unable/unwilling to undergo cessation of oral antihistamines for five days prior to testing.
* Current use of oral steroids or other systemic immunosuppressants, including omalizumab (anti-IgE therapy) and anti-IL-5 therapy.
* Allergic asthmatics with current uncontrolled asthma.
* Pregnant women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-05-15 (Actual); Primary Completion 2022-05-14 (Estimated); Study Completion 2022-05-14 (Estimated)

PRIMARY OUTCOMES:
Change in Mean Allergen Induced Wheal Diameter | 60 minutes
  Greatest diameter millimeters and orthogonal diameter millimeters, mean of both

CONTACTS AND LOCATIONS:
Overall Officials: Rauno O Joks, MD, Principal Investigator — State University of New York - Downstate Medical Center
Locations (1):
- SUNY Downstate Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No
No plan.